CLINICAL TRIAL: NCT01656148
Title: Fampyra Outcome Measures Study: a Study of Different Outcome Measures on the Effect of Fampyra
Brief Title: FAME - Fampyra Outcome Measures Study: a Study of Different Outcome Measures on the Effect of Fampyra
Acronym: FAME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); Biogen (Industry)
Responsible Party: Principal Investigator, Henrik Boye Jensen, MD, PhD Fellow, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FAME; 2011-006151-10 (EudraCT Number)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Walking disablility; Mobility; Six Spot Step Test; Outcome measures; Fampridine-SR; Fampyra
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fampridine-SR (Experimental): Initially all participants receive Fampridine-SR 10 mg BID in an open label enrichment phase lasting four weeks. Those 40% responding the most by SSST will go onto phase two. 50% of these will receive 10 mg Fampridine-SR BID for four weeks.
  Interventions: Drug: Fampridine-SR
- Placebo (Placebo Comparator): In the intervention phase 50% will receive placebo BID
  Interventions: Drug: Fampridine-SR

INTERVENTIONS:
Drug: Fampridine-SR — Subjects will all receive Fampridine-SR in an open label enrichment phase lasting four weeks. Those 40% improvin the most measured by SSST will go onto the intervention. Here randomization in a 1:1 key between Fampridine-SR and placebo will be undertaken. Treatment will be of either Fampridine-SR 10 mg BID or placebo BID for four weeks. Arms will be double blind.
  Other Names: Fampyra (Ampyra in the US).

SUMMARY:
Fampridine-SR is registered for the treatment of walking incapacity in MS patients. Two pivotal trials show that app. 40% of MS patients with walking incapacity can improve walking speed averagely 25% when recieving the drug. This has been shown using the Timed 25 Foot Walk Test (T25FW). No effect on cognition and upper limb function has been shown, but this has not been investigated in patients responding to the drug measured by the abovementioned test.

The question is if this will be the case and also if another walking test, termed the Six Spot Step Test (SSST), will be more sensitive to the effect of Fampridine-SR.

Primary outcome measure is the effect measured by SSST. The hypothesis is that SSST is not less sensitive to the effect of Fampridine-SR than T25FW.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically definite multiple sclerosis diagnosed according to the McDonald criteria
* EDSS 4-7
* Pyramidal FS >= 2

Exclusion Criteria:

* History of epileptic seizures
* MS relapse or change in disease modifying treatment (DMT) within 60 days
* cancer within five years
* uncontrolled hypertension
* clinically important cardiac, hepatic, renal or pulmonary disease
* pregnancy
* breast feeding
* concomitant treatment with cimetidine, carvedilol, propranolol and metformin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The mean change in SSST | SSST is measured before and at the end of four weeks of treatment
  SSST is measured before treatment with Fampridine-SR. Then again measured at day 26, 27 or 28 of four weeks of treatment with Fampridine-SR.

SECONDARY OUTCOMES:
Mean change in T25FW | Four weeks
  T25FW is measured before four weeks of treatment with Fampridine-SR and then on day 26, 27 or 28.
Mean change in hip flexion, knee flexion and knee extension force | Four weeks
  Force in the abovementioned areas is measured by dynamometry before four weeks of treatment with Fampridine-SR and on day 26, 27 or 28.
Mean change on Chair Rise Test | Four weeks
  Time to rise from a chair five times is measured before four weeks of treatment with Fampridine-SR and on day 26, 27 or 28.
Mean change on 9-Hole Peg Test (9HPT) | Four weeks
  9HPT is measured before four weeks of treatment with Fampridine-SR and on day 26, 27 or 28.
Mean change on Symbol Digit Modalitites Test (SDMT) | Four weeks
  SDMT is measured before four weeks of treatment with Fampridine-SR and on day 26, 27 or 28.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik B Jensen, MD, Principal Investigator — Institute for Regional Health Services Research, University of Southern Denmark
Locations (4):
- Denmark (4):
  - Esbjerg Hospital, Esbjerg
  - Odense University Hospital, Odense
  - Sønderborg Hospital, Sønderborg
  - Vejle Hospital, Vejle

REFERENCES:
- [Background] Solari A, Uitdehaag B, Giuliani G, Pucci E, Taus C. Aminopyridines for symptomatic treatment in multiple sclerosis. Cochrane Database Syst Rev. 2002;(4):CD001330. doi: 10.1002/14651858.CD001330. PMID 12804404
- [Background] Judge SI, Bever CT Jr. Potassium channel blockers in multiple sclerosis: neuronal Kv channels and effects of symptomatic treatment. Pharmacol Ther. 2006 Jul;111(1):224-59. doi: 10.1016/j.pharmthera.2005.10.006. Epub 2006 Feb 9. PMID 16472864
- [Background] Schwid SR, Petrie MD, McDermott MP, Tierney DS, Mason DH, Goodman AD. Quantitative assessment of sustained-release 4-aminopyridine for symptomatic treatment of multiple sclerosis. Neurology. 1997 Apr;48(4):817-21. doi: 10.1212/wnl.48.4.817. PMID 9109861
- [Background] Goodman AD, Cohen JA, Cross A, Vollmer T, Rizzo M, Cohen R, Marinucci L, Blight AR. Fampridine-SR in multiple sclerosis: a randomized, double-blind, placebo-controlled, dose-ranging study. Mult Scler. 2007 Apr;13(3):357-68. doi: 10.1177/1352458506069538. Epub 2007 Jan 29. PMID 17439905
- [Background] Goodman AD, Brown TR, Krupp LB, Schapiro RT, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F203 Investigators. Sustained-release oral fampridine in multiple sclerosis: a randomised, double-blind, controlled trial. Lancet. 2009 Feb 28;373(9665):732-8. doi: 10.1016/S0140-6736(09)60442-6. PMID 19249634
- [Background] Goodman AD, Brown TR, Cohen JA, Krupp LB, Schapiro R, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F202 Study Group. Dose comparison trial of sustained-release fampridine in multiple sclerosis. Neurology. 2008 Oct 7;71(15):1134-41. doi: 10.1212/01.wnl.0000326213.89576.0e. Epub 2008 Jul 30. PMID 18672472
- [Background] Goodman AD, Brown TR, Edwards KR, Krupp LB, Schapiro RT, Cohen R, Marinucci LN, Blight AR; MSF204 Investigators. A phase 3 trial of extended release oral dalfampridine in multiple sclerosis. Ann Neurol. 2010 Oct;68(4):494-502. doi: 10.1002/ana.22240. PMID 20976768
- [Background] Cutter GR, Baier ML, Rudick RA, Cookfair DL, Fischer JS, Petkau J, Syndulko K, Weinshenker BG, Antel JP, Confavreux C, Ellison GW, Lublin F, Miller AE, Rao SM, Reingold S, Thompson A, Willoughby E. Development of a multiple sclerosis functional composite as a clinical trial outcome measure. Brain. 1999 May;122 ( Pt 5):871-82. doi: 10.1093/brain/122.5.871. PMID 10355672
- [Background] Nieuwenhuis MM, Van Tongeren H, Sorensen PS, Ravnborg M. The six spot step test: a new measurement for walking ability in multiple sclerosis. Mult Scler. 2006 Aug;12(4):495-500. doi: 10.1191/1352458506ms1293oa. PMID 16900764
- [Derived] Jensen HB, Nielsen JL, Ravnborg M, Dalgas U, Aagaard P, Stenager E. Effect of slow release-Fampridine on muscle strength, rate of force development, functional capacity and cognitive function in an enriched population of MS patients. A randomized, double blind, placebo controlled study. Mult Scler Relat Disord. 2016 Nov;10:137-144. doi: 10.1016/j.msard.2016.07.019. Epub 2016 Sep 14. PMID 27919481
- [Derived] Jensen H, Ravnborg M, Mamoei S, Dalgas U, Stenager E. Changes in cognition, arm function and lower body function after slow-release Fampridine treatment. Mult Scler. 2014 Dec;20(14):1872-80. doi: 10.1177/1352458514533844. Epub 2014 May 22. PMID 24852920